CLINICAL TRIAL: NCT02449265
Title: Efficacy of Consolidative Involved-site Radiotherapy Following Sufficient Chemotherapy for Patients With Limited-stage Diffuse Large B-cell Lymphoma: Wuhan University Cancer Center -NHL03 Trial
Brief Title: Efficacy of Consolidative Involved-site Radiotherapy for Patients With Limited-stage Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Di Deng, Director, Clinical Research, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUCC-NHL03 Trial
Record Dates: First submitted 2015-05-07; First posted 2015-05-20 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: limited-stage DLBCL; consolidation involved-site radiotherapy; Chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ISRT group (Experimental): Six cycles chemotherapy (cyclophosphamide 750mg/square meter on day 1 + doxorubicin 50mg/square meter on day 1 + vincristine 1.4mg/square meter on day 1 (up to a maximal dose of 2 mg) +prednisone 60mg/square meter on day 1 through 5, repeated at 21-day intervals).
  Consolidation involved-site radiotherapy (ISRT) following in patients with complete or paratial response beginning 1 month after the last cycle of chemotherapy.
  Interventions: Radiation: Consolidation involved-site radiotherapy (ISRT); Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone
- IFRT group (Active Comparator): Six cycles chemotherapy (cyclophosphamide 750mg/square meter on day 1 + doxorubicin 50mg/square meter on day 1 + vincristine 1.4mg/square meter on day 1 (up to a maximal dose of 2 mg) +prednisone 60mg/square meter on day 1 through 5,repeated at 21-day intervals ).
  Consolidation involved-field radiotherapy (IFRT) following in patients with complete or paratial response beginning 1 month after the last cycle of chemotherapy.
  Interventions: Radiation: Consolidation involved-field radiotherapy (IFRT); Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone

INTERVENTIONS:
Radiation: Consolidation involved-site radiotherapy (ISRT) — 6 cycles modern CHOP chemotherapy. Involved-site radiotherapy (ISRT) is based on defining the site of gross disease before chemotherapy, the GTV and using a CT-based volume with an expansion to form a CTV in the cranio-caudal direction.
  The general dose had been guided that 30-36Gy in 15~18 fractions of 2 Gy 5 days per week was managed for patients with complete response (CR) after chemotherapy and 40-50Gy in 20~25 fractions of 2 Gy 5 days per week for partial response (PR).
  Arms: ISRT group
Radiation: Consolidation involved-field radiotherapy (IFRT) — 6 cycles modern CHOP chemotherapy. Radiotherapy field of IFRT defined by CALGB is encompassed the prechemotherapy gross tumor.
  The general dose had been guided that 30-36Gy in 15~18 fractions of 2 Gy 5 days per week was managed for patients with complete response (CR) after chemotherapy and 40-50Gy in 15~18 fractions of 2 Gy 5 days per week for partial response (PR).
  Arms: IFRT group
Drug: cyclophosphamide — Patients in both arms will be given cyclophpsphamide chemotherapy.
Drug: doxorubicin — Patients in both arms will be given doxorubicin chemotherapy.
Drug: vincristine — Patients in both arms will be given vincristine chemotherapy.
Drug: prednisone — Patients in both arms will be given prednisone chemotherapy.

SUMMARY:
The most common option of radiotherapy for patients with limited-stage DLBCL is involved-field radiotherapy (IFRT). The more limited radiotherapy field size changing from IFRT to reasonable margin from gross tumor has been reported to maintain the high rates of local disease control, while minimizing the risks of radiation-induced toxicities. However, the research didn't analyze whether the efficacy of consolidation involved-site radiotherapy (ISRT) be affected by the response of chemotherapy. The biologic definition of clinical target volume (CTV) of ISRT and actual radiotherapy field size need to be ascertained.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is a heterogenous group of lymphomas and constitutes approximately one-third of all non-Hodgkin lymphoma diagnoses. At diagnosis, approximately 25% to 30% of patients are found to have limited-stage disease (stage I-II). The combined-modality therapy (CMT) including chemotherapy and involved-field radiotherapy (IFRT) is the optimal management of limited-stage DLBCL. The National Comprehensive Cancer Network (NCCN) guidelines recommend three cycles of R-CHOP+IFRT for early-stage, nonbulky disease but also allow the administration of six to eight cycles of R-CHOP with or without IFRT. These patients have a favorable prognosis with 5-year overall survival (OS) rates reported between 70% and 92% following curative-intent treatments.

In fact, the value from consolidation radiotherapy (RT) in limited-stage DLBCL is uncertain in several well-known reports. These include the report of late relapses in the SWOG study, the lack of benefit for adding RT to brief chemotherapy in a European study of elderly patients, and the reported advantage of an intensive chemotherapy regimen over brief CHOP plus RT in younger patients studied in Europe. On the other hand, it is uncertain how many cycles' chemotherapy combining consolidation RT is adequate to maintain the efficacy of CMT for patients with limited-stage DLBCL. In the trial of GELA LNH 93-1, an aggressive chemotherapy alone, a regimen were dose-intensified doxorubicin, cyclophosphamide, vindesine, bleomycin, and prednisone (ACVBP), was designed to compare with three cycles of CHOP plus IFRT in patients with stage I-II mostly low-risk aggressive lymphoma. Patients who receive the dose-intensity chemotherapy had significantly higher 5-year event-free and overall survival (OS) rates because the abbreviated therapy was not enough to overcome the excessive distant relapses. In the SWOG 8736 trial, the results were clearly in favor of keeping RT on board, but the progression-free survival (PFS) and OS curves between three cycles of CHOP+IFRT arm and eight cycles of CHOP arm begin to overlap at 7 years and at 9 years after treatment because of the excess number of late lymphoma relapses in the group that received three cycles of CHOP+IFRT. For patients older than 60 years with localized aggressive lymphoma, the results of the GELA LNH 93-4 trial show that 5-year event-free survival (EFS) and OS were no significant differences between four cycles of CHOP alone and four cycles of CHOP followed by radiation therapy. In summary, it is not sufficient that three cycles of CHOP as systemic treatment in the abbreviated therapy treated limited-stage DLBCL according to the results of previous randomized trials. These findings are consistent with the retrospective results of the M. D. Anderson Cancer Center (MDACC). Six to eight cycles of chemotherapy may be the adequate management for patients with limited-stage DLBCL who received RT to ensure a significantly better outcome.

In order to increase the clinical benefit and decrease the late complications related to irradiation and/or chemotherapy, consolidation RT following chemotherapy in patients with limited-stage DLBCL has been directed in recent years. This is based on the observation that local recurrence is the most common pattern of first failure following systemic therapy alone and IFRT achieves excellent infield control in the original sites of disease. Improved local control, achieved by the addition of radiotherapy, may translate into improvements in long-term outcomes. The advantages of the addition of RT are obvious in the reduction of adverse events of dose-intensified or more cycles' chemotherapy, in the increase of local control, and even in the improvement of OS. However, the complications related to consolidation RT, including second malignancies and other non-neoplastic late events, were also needed to emphasize for those patients with limited-stage DLBCL, who were cured and have a long-term survival. Reducing the morbidity of treatment is an important consideration to optimize the therapeutic ratio. The prefer options include radiation field size reduction and radiotherapy dose decrease. The general dose had been guided that 30-36Gy was managed for patients with complete response (CR) after chemotherapy and 40-50Gy for partial response (PR). Comparing to extensive-field radiotherapy, the brief chemotherapy followed by IFRT for early-stage disease is safe and significantly more effective. In order to maintain the high rates of local disease control achieved by RT, while minimizing the risks of radiation-induced toxicities, the more limited radiotherapy field size changing from IFRT to reasonable margin from gross tumor has been reported in patients with limited-stage DLBCL. The Korean retrospective results reported by Yu show that the OS and relapse-free survival (RFS) at 10 years managed by Involved-node radiotherapy (INRT) following median 4 cycles of CHOP or R-CHOP chemotherapy has the same treatment results compared to IFRT on 86 patients with stage I, II head and neck DLBCL. The radiotherapy field size of INRT are more localized to cover the prechemotherapy gross disease with margins of at least 2 to 3 cm while not include ipsilateral whole neck. Aim to reduce radiotherapy-induced toxicities, Campbell et al. reduced the field size from IFRT to INRT<5 cm in the treatment of limited-stage DLBCL with abbreviated systemic therapy and consolidation RT. The results show that distant-only relapse was the most common pattern of first failure, and marginal-only relapse was reassuringly infrequent (2%) in the group of INRT. The TTP, PFS, and OS don't be affected by radiotherapy field reduction.

Smaller RT fields will translate to lower rates of radiation-induced toxicity and radiation-induced second malignancy in long-term survivors. Unfortunately, some limitation of the INRT reported in previous studies will be undertaken. The involved sites are only in head and neck and comparison arms are not designed in the Korean research. Though the results of Campbell et al show that reducing the field size from IFRT to INRT<5 cm maintains a low marginal recurrence risk with no impact on overall outcome, the research was retrospective and didn't analyze whether the efficacy of consolidation INRT be affected by the response of chemotherapy. Moreover, the clinical target volume (CTV) of INRT in the research of Campbell et al encompassed the prechemotherapy volume of disease, within postchemotherapy anatomical limits instead of biologic region of the subclinical of gross disease. At the same time, a physical concept, the planning target volume (PTV) must be formed from CTV considering physiological movement and interfraction set-up variation. For this, the up-to 5 cm directed in "involved-node radiotherapy with margins up to 5 cm (INRT<5 cm) '' by Campbell et al accounts for the non-uniform margins. The actual radiotherapy field size varied according to the discretion of the treating radiation oncologist.

It is necessary that a research without the limitation being in previous study should be designed to evaluate the efficacy of RT with smaller RT field size following sufficient systemic treatment for patients with limited-stage DLBCL. Involved-site radiotherapy (ISRT), based on a modified involved field, aims to reduce the radiation volume treated and the probability of late effects. Its radiation targets include a gross tumor volume (GTV), a clinical target volume (CTV), and a planning target volume (PTV), which were defined in International Commission on Radiation Units and Measurements Report (ICRU) 50. This is based on defining the site of gross disease before chemotherapy, the GTV and using a CT-based volume with an expansion to form a CTV in the cranio-caudal direction.

Compared to the IFRT, the PFS and toxicities related to involved-site radiotherapy (ISRT) were to be evaluated for CR and PR patients with limited-stage DLBCL after sufficient systemic treatment. The CTV of ISRT is defined as the region including the prechemotherapy volume of disease with 1.5 cm margin expanded cranio-caudally in the direction of potential lymphatic spread. The CTV should not extend into air in the transverse plane and should be limited in the involved lymph node region defined by the Cancer and Leukemia Group B (CALGB). The PTV is then extended from CTV by adding the necessary margin for setup error and organ motion.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female aged range from 18 years to 65 years.
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1.
* All patients had histologically confirmed Diffuse large B-cell lymphoma.
* Limited-stage DLBCL patients at newly diagnosed or recurrent without RT in initial management.
* Adequate organ function.
* Negative pregnancy test.
* Signed informed consent document on file.

Exclusion Criteria:

* Woman who were pregnant or lactating.
* With severe local infection or general infective disease.
* Primary lymphoma in special organ including cuticula, center never system, gastrointestinal tract, testicle, and lung.
* With other second primary malignancy except cutaneum carcinoma.
* Being or planning to participate in other study.
* Any patient who in the opinion of the investigator should not participate in the study.

Withdrawal Criteria:

* Patient are free to withdrawal completely from the study at any time upon request.
* Patient in the study may be stopped with the patient agreement at any time at the discretion of investigator.
* In-field progression on irradiation ongoing.
* Poor tolerability adverse events in the period of chemotherapy or irradiation after enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival - PFS | from the date of diagnosis to the date of treatment failure or death from any cause, whichever occurs first, Assessed up to 100 months.
  Treatment failure was defined as any recurrence of non-Hodgkin lymphoma.
Adverse events with grade 3 or 4 - AEs | The time from the day of treatment to the day of the first documented disease progression or death from any cause, Assessed up to 24 months.
  Toxicity was scored according to the toxicity scale of the National Cancer Institute Common Terminology Criteria for Adverse Events 3.0.

SECONDARY OUTCOMES:
Overall survival - OS | Time Frame: From the initial diagnosis of follicular lymphoma to death from any cause, Assessed up to 120 months.
Rate of in-field progression | From the start of RT to the first documented disease progression within the radiotherapy field, Assessed up to 100 months.
Rate of out-field progression | From the start of RT to the first documented disease progression outside the radiotherapy field, Assessed up to 100 months.
Rate of regional failure | From the start of RT to the first documented disease progression outside of ISRT field but within the involved region defined as CALGB, Assessed up to 100 months.

CONTACTS AND LOCATIONS:
Locations (1):
- DiDeng, Wuhan, Hubei, China